CLINICAL TRIAL: NCT02349438
Title: Assessment of Contact Lens Wettability Using Wavefront Aberrometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CR-5685
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A (Experimental): The lenses will be worn for 2 hours in both eyes, and not dispensed
  Interventions: Device: senofilcon A; Device: lotrafilcon B
- lotrafilcon A (Active Comparator): The lenses will be worn for 2 hours in both eyes, and not dispensed
  Interventions: Device: senofilcon A; Device: lotrafilcon B

INTERVENTIONS:
Device: senofilcon A — A soft spherical contact lens
Device: lotrafilcon B

SUMMARY:
This study will test the feasibility that differences in contact lens wettability can be measured with a wavefront sensor.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or females that are at least 18 to no more than 40 years of age.
2. The subject must read, understand, and sign the Statement of Informed Consent and receive a fully executed copy of the form.
3. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
4. The subject must possess a wearable pair of spectacles with distance vision correction which provide satisfactory vision.
5. The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of lens wear per week for a minimum of 1 month prior to the study) or has sufficient prior experience with soft contact lens wear (defined as a minimum of 30 days of lens wear during the last 5 years).
6. The subject's vertexed best sphere distance refraction must be between -0.75 and -5.00 D in both eyes.
7. Cylinder refraction less than or equal to -0.75 D in both eyes (any axis).
8. The subject must have corrected visual acuity of 20/20 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
4. Any known hypersensitivity or allergic reaction to contact lens solutions or sodium fluorescein dye.
5. Any previous ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.)
6. Current wearers of rigid or hybrid contact lenses.
7. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion by keratometry.
8. Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
9. History of binocular vision abnormality or strabismus.
10. Employee of the investigational clinic (e.g. Investigator, Coordinator, Technician).
11. Clinically significant (grade 3 or 4) corneal edema, pterygium, corneal vascularization, corneal staining, or any other abnormalities of the cornea or conjunctiva which may interfere with the study measurements.
12. Strabismus, suppression or amblyopia.
13. Any ocular infection.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kelvin Grove, Queensland, Australia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 25 subjects were enrolled into this study. Of the enrolled subjects 4 did not meet the eligibility criteria and 21 were dispensed study lenses. Of the dispensed subjects all 21 completed the study.
Groups:
- Senofilcon A/Lotrafilcon B: Subjects that were randomized to receive the senofilcon A lens first and then to receive the lotrafilcon B lens.
- Lotrafilcon B/Senofilcon A: Subjects that were randomized to receive the lotrafilcon B lens first and then to receive the senofilcon A lens.
Period: Period 1
Arm/Group | Senofilcon A/Lotrafilcon B | Lotrafilcon B/Senofilcon A
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Senofilcon A/Lotrafilcon B | Lotrafilcon B/Senofilcon A
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed at least 1 study lens throughout the duration of the study.
Groups:
- Dispensed: All subjects that were dispensed at least 1 study lens during the course of the study.
Arm/Group | Dispensed
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.1 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 14
  White | 7
Region of Enrollment [Number; unit: participants]
  Australia | 21

OUTCOME MEASURES:

1. Primary Outcome: Higher Order Root Mean Square (HO RMS) - Near Target in Downgaze With Natural Blinking
Description: Wavefront metric measured by COAS wavefront sensor while subject fixates a near digital device in a down-gaze position with natural blinking. The average HO RMS was reported for each lens. Lower values indicate better outcome.
Time Frame: 2 hours post insertion
Population: All subjects that have completed all study visits.
Measure: Mean (Standard Deviation); unit: microns
Groups:
- Senofilcon A: Subjects that wore the senofilcon A lens in either the 1st or 2nd period of the study.
- Lotrafilcon B: Subject that wore the lotrafilcon B in either the 1st or 2nd period of the study.
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 21 | 21
microns | 0.159 (0.0662) | 0.142 (0.0605)

2. Primary Outcome: Higher Order Root Mean Square (HO RMS) - Near Target in Downgaze With Controlled Blink
Description: Wavefront metric measured by COAS wavefront sensor while subject fixates a near digital device in a down-gaze position with controlled blinking. The average HO RMS was reported for each lens. Lower values indicate better outcome.
Time Frame: 2 hours post insertion
Population: All subjects that have completed all study visits.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 21 | 21
microns | 0.165 (0.0857) | 0.146 (0.0567)

3. Primary Outcome: Higher Order Root Mean Square (HO RMS) - Distance Target in Primary Gaze With Controlled Blink
Description: Wavefront metric measured by COAS wavefront sensor while subject fixates a distant target in primary gaze with controlled blinking. The average HO RMS was reported for each lens. Lower values indicate better outcome.
Time Frame: 2 hours post insertion
Population: All subjects that have completed all study visits.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Senofilcon A | Lotrafilcon B
Number analyzed (Participants) | 21 | 21
microns | 0.125 (0.0559) | 0.132 (0.0511)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1-week per subject.
Arm/Group | Senofilcon A | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days